CLINICAL TRIAL: NCT04753671
Title: Normal Pregnancy and Postpartum Reference Ranges Intervals for QUANTRA® (STAGO BIOCARE) Hemostasis Point of Care Device
Brief Title: QUANTRA® References Range Protocol in Pregnancy and Postpartum
Acronym: QUANTRA®_GPP
Status: Completed | Type: Observational
Sponsor: University Hospital, Lille (Other)
Responsible Party: Sponsor
Other Study IDs: 2020_14; 2020-A03000-39 (Other: ID-RCB number,ANSM)
Record Dates: First submitted 2021-02-08; First posted 2021-02-15 (Actual); Last update posted 2025-12-26 (Actual); Status verified 2025-12

CONDITIONS: Pregnancy Postpartum
Keywords: Hemostasis; pregnancy; postpartum; point of care; coagulopathy
MeSH Terms: conditions — Hemostatic Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Postpartum hemorrhage (PPH) remains the leading cause of maternal death. PPH associated coagulopathy varies and their treatments (tranexamic acid, fibrinogen concentrates,plasma, platelets need to be targeted and administrated early. Point of care hemostasis devices are helpful to develop this strategy. Quantra® (STAGO BIOCARE) use an innovative method to detect the clot formation. Pregnancy and non-hemorrhagic postpartum reference ranges are missing. The objective of this study is to establish these norms needed to elaborate thereafter the thresholds to be targeted in PPH conditions.

ELIGIBILITY:
Inclusion Criteria:

* Healthy pregnant woman (indemne of any chronic pathology neither obstetrical pathology)
* Delivering vaginally without postpartum hemorrhage for 60 patients
* Delivering through a programmed C-section for 20 patients
* Having given a non-opposition agreement to participate in the study.
* Major patient with social insurance

Exclusion Criteria:

* Any acute or chronic hemostasis pathology before pregnancy or during pregnancy instrumental delivery or cesarean section Postpartum bleeding.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — pregnant women
Study Population: a cohort of Healthy pregnant woman (indemne of any chronic pathology neither obstetrical pathology)
Sampling Method: Probability Sample
Enrollment: 31 (Actual)
Dates: Start 2021-05-05 (Actual); Primary Completion 2022-11-07 (Actual); Study Completion 2022-11-07 (Actual)

PRIMARY OUTCOMES:
Description of the QUANTRA® parameters range intervals before and after vaginal delivery | At admission (= before delivery )
Description of the QUANTRA® parameters range intervals before and after vaginal delivery | At 30 minutes +/- 10 minutes after delivery

SECONDARY OUTCOMES:
Description of the QUANTRA® parameters range intervals before and after vaginal delivery | At 30 up to 60 minutes after birth and placental removal.
Comparison between end of pregnancy and immediate postpartum reference values (both vaginal and caesarean deliveries) | At 30 up to 60 minutes after birth

CONTACTS AND LOCATIONS:
Overall Officials: Anne-Sophie DUCLOY-BOUTHORS, MD, Principal Investigator — University Hospital, Lille
Locations (1):
- Hop Jeanne de Flandre Chu Lille, Lille, France

REFERENCES:
- [Result] Lukowiak O, Le Gouez A, Djebbour M, Mercier FJ, Bouthors AS. Peri-partum reference range for the point-of-care viscoelastic testing device Quantra(R) QStat in healthy pregnancy and non-haemorrhagic post-partum - A short communication. Anaesth Crit Care Pain Med. 2025 Aug;44(4):101521. doi: 10.1016/j.accpm.2025.101521. Epub 2025 Apr 17. PMID 40252700